CLINICAL TRIAL: NCT05404503
Title: Analysis of the Incidence of Cholangiocarcinoma on Choledochal Cyst in a Western Center
Acronym: QuiCo
Status: Enrolling by invitation | Type: Observational
Sponsor: María Teresa Moreno Asencio (Other)
Responsible Party: Principal Investigator, María Teresa Moreno Asencio, MorenoAsencioM, Fundación Andaluza Beturia para la Investigación en Salud
Other Study IDs: MorenoAsencioM
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Incidence of Cholangiocarcinoma on Choledochal Cysts; Postoperative Complications in Choledochal Cysts; Choledochal Cyst Monitoring
Keywords: cholangiocarcinoma, choledochal cysts, surgery
MeSH Terms: conditions — Cholangiocarcinoma; Choledochal Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Choledochal cysts are congenital cystic dilatations of the intra and/or extrahepatic bile duct. They have been considered a rare entity of the child population. Globally, they account for 1% of all biliary pathology benign, with a clearly higher incidence in Asian countries (1/5,000 in China, 1/1,000 in Japan, compared to 1/100,000-150,000 in Western countries). However, the number of adults diagnosed in recent years has increased by up to 70% due to improvements in imaging tests.

Currently, the common bile duct malformation is considered a premalignant entity: although the data are not very precise, it is estimated that between 2.6% and 26% of patients diagnosed choledochal cyst, will develop cholangiocarcinoma. In this sense, we must bear in mind that most of the published literature is of Asian origin, where the rate of cholangiocarcinoma is 0.1-71/100,000 compared to 0.1-1.8/100,000 in Europe or 0.6-1/100,000 in the USA.

The most used classification to differentiate the types of cysts is that of Todani. Following this classification, we would find a higher rate of malignancy on types I and IV.

The recommendations found in the literature refer to the need for surgical intervention for choledochal cysts due to their high rate of malignancy. These recommendations are based on studies conducted in a symptomatic Asian population. We do not usually find in therapeutic algorithms the inclusion of various factors that could be involved in the development of malignancy such as episodes of cholangitis, presence of anomaly in the pancreatobiliary junction, presence of lithiasis in cystic dilatation, etc.

Some surveys carried out among the scientific population reflect a lack of consensus on its management: in the same clinical situation, different surgery units specialized in hepatobiliary-pancreatic pathology would act in the opposite way (specifically surgical versus conservative treatment).

Bile duct resection is not without complications, both short-term and long-term. Therefore, the patient's symptoms, age or comorbidities can play an important role in decision-making in the treatment of this pathology.

This nationwide multicenter retrospective observational study aims to determine the clinical situation of this rare pathology in a Western environment.

A retrospective analysis of patients diagnosed with choledochal cyst in the period between 2000 and 2020 is proposed. Demographic variables, risk factors for cholangiocarcinoma, symptoms associated with the cyst and its characteristics, diagnostic method, type of treatment, complications will be analyzed. Malignancy, time, and follow-up method will also be discussed.

This study will attempt to answer questions about the incidence of choledochal cysts in our environment, their association with cholangiocarcinoma, the associated morbidity and mortality, as well as the therapeutic and follow-up attitudes adopted in the face of this rare pathology.

ELIGIBILITY:
Inclusion Criteria:

- A radiological diagnosis (diagnosed by the radiology service) of choledochal cyst, understood as a dilatation of the extra or intrahepatic bile duct (fusiform or saccular, following the Todani classification)

Exclusion Criteria:

* An objectified obstructive cause that justifies a dilatación of bile duct (lithiasis, papillitis or neoplasia)
* A definitive imaging test that rules out an initial diagnosis of choledochal cyst.
* Intraoperative diagnosis of choledochal cyst without subsequent radiological confirmation.
* Patients with cystic lesions of another nature (biliary cysts, simple cysts, cystic neoplasms).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a radiological diagnosis of choledochal cyst. Those patients diagnosed by the radiology service are included
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Choledochal cyst and cholangiocarcinoma | 20 years
  to analyze the incidence of cholangiocarcinoma in choledochal cysts

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Ramón Jimenez Hospital, Huelva, Spain